

# Non-Interventional Study (NIS) Protocol

| | 25044226.04 |
|---|---|
| Document Number: | c37044336-01 |
| BI Study Number: | 1160-0308 |
| BI Investigational Product(s): | Pradaxa |
| Title: | Comparative safety and effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD) |
| Brief lay title: | A study based on Japanese medical records that looks at bleeding events in people with atrial fibrillation and coronary artery disease who start taking either dabigatran, rivaroxaban, or warfarin |
| Protocol version identifier: | 1.0 |
| Date of last version of protocol: | Not applicable |
| PASS: | Yes |
| EU PAS register number: | EUPAS41345 |
| Active substance: | Dabigatran, warfarin, rivaroxaban |
| Medicinal product: | Pradaxa, Xarelto |
| Product reference: | 1160 |
| Procedure number: | Not applicable |
| Marketing authorisation holder(s): | |
| Joint PASS: | No |
| Research question and objectives: | The study aims to evaluate the safety and effectiveness comparisons between warfarin, dabigatran, and rivaroxaban in routine clinical practice among Japanese NVAF patients with concomitant CAD. |
| | Primary objective: |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| | To compare the risk of major bleeding between dabigatran and warfarin, and between rivaroxaban and warfarin, among Japanese NVAF patients with concomitant CAD. |
|---|---|
| | Secondary objective: To compare the net clinical benefits of dabigatran vs. warfarin, and rivaroxaban vs. warfarin, among Japanese NVAF patients with concomitant CAD. |
| | Further objective: If the required sample size can be fulfilled and the baseline characteristics are balanced between dabigatran and rivaroxaban groups after IPTW adjustment, to compare the safety and net clinical benefits of dabigatran vs rivaroxaban among Japanese NVAF patients with concomitant CAD. |
| Country(-ies) of study: | Japan |
| Author: | Observational Study Specialist, |
| Marketing authorisation holder(s): | |
| | Phone: Fax: |
| In case of PASS, add: MAH contact person: | |
| In case of PASS, add:<br><eu-qppv:></eu-qppv:> | Phone: Fax: 24-hour phone contact: |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| In case of PASS, add: <signature eu-="" of="" qppv:=""></signature> | |
|---|---|
| Date: | 15 Nov 2021 |
| Proprietary confidential information © 2021 Boehringer Ingelheim Group of companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission | |

## NIS Protocol BI Study Number 1160-0308

 c37044336-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 1. TABLE OF CONTENTS

| TITLE | PAGE | | 1 |
|-------|----------|--------------------------------|----|
| 1. T | ABLE O | F CONTENTS | 4 |
| 2. L | IST OF A | ABBREVIATIONS | 6 |
| 3. R | ESPONS | SIBLE PARTIES | 8 |
| 4. A | BSTRAG | CT | 9 |
| 5. A | MENDN | MENTS AND UPDATES | 17 |
| 6. N | ILESTO | ONES | 18 |
| 7. R | ATIONA | ALE AND BACKGROUND | 18 |
| 8. R | ESEARO | CH QUESTION AND OBJECTIVES | 19 |
| 9. R | ESEARO | CH METHODS | 19 |
| 9.1 | STUDY | Y DESIGN | 19 |
| 9.2 | SETTI | NG | 20 |
| 9.2 | .1 Str | udy Sites | 20 |
| 9.2 | .2 Str | udy population | 21 |
| 9.2 | .3 Str | udy visits | 21 |
| 9.2 | .4 Str | udy discontinuation | 21 |
| 9.3 | VARIA | ABLES | 21 |
| 9.3 | .1 Ex | xposures | 21 |
| 9.3 | .2 Ou | utcomes | 22 |
| 9 | 0.3.2.1 | Primary outcomes | |
| 9 | 0.3.2.2 | Secondary outcomes | 22 |
| 9.3 | | ovariates | |
| 9.4 | | SOURCES | |
| 9.5 | | Y SIZE | |
| 9.6 | | MANAGEMENT | |
| 9.7 | | ANALYSIS | |
| 9.7 | .1 Ma | ain analysis | 25 |
| 9.7 | | Ifety Analysis | |
| 9.8 | | ITY CONTROL | |
| 9.9 | | ATIONS OF THE RESEARCH METHODS | |
| 9.10 | OTHE | R ASPECTS | 27 |

## NIS Protocol BI Study Number 1160-0308

 **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Data quality assurance 27 9.10.1 9.10.2 Study records 27 9.10.2.1 9.10.2.2 Protocol deviations 28 9.10.3 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED 10.2 MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS 28 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND 11.1 11.2 PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS 29 13. ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES ...... 45

**NIS Protocol** BI Study Number 1160-0308

 c37044336-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

ADR Adverse Drug Reaction

AΕ Adverse Event Atrial Fibrillation AF

**ASD** Absolute Standardized Difference

Competent Authority CA CAD Coronary Artery Disease CCDS Company Core Data Sheet

CHA2DS2-Congestive heart failure, Hypertension, Age ≥ 75 years, Diabetes **VASc** 

mellitus, Stroke, Vascular disease, Age 65-74 years, Sex category

(female)

Confidence Interval CI **CML** Local Clinical Monitor **CRA** Clinical Research Associate

**CRF** Case Report Form CTP Clinical Trial Protocol

**DMRP** Data Management and Review Plan

**Electronic Case Report Form eCRF** 

**ENCePP** European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

European Medicines Agency **EMA** European Society of Cardiology **ESC** Food and Drug Administration **FDA** 

Good Clinical Practice **GCP** 

Good Epidemiological Practice **GEP** 

Gastrointestinal GI

**GPP** Good Pharmacoepidemiology Practice **GVP** Good Pharmacovigilance Practices

Hypertension, Abnormal renal/liver function, Stroke, Bleeding history or **HAS-BLED** 

predisposition, Labile INR, Elderly (>65 years), Drugs/alcohol

concomitantly

Hazard Ratio HR

ΙB Investigator's Brochure

The 10<sup>th</sup> Revision of the International Classification of Diseases ICD-10

Intracranial Hemorrhage **ICH** ID **Identification Number** 

**Independent Ethics Committee IEC** 

**IPTW** Inverse Probability of Treatment Weighting

**IRB** Institutional Review Board MAH Marketing Authorization Holder

MedDRA Medical Dictionary for Regulatory Activities

Myocardial Infarction MI Non-Interventional Study **NIS** 

Non-vitamin K Oral Anticoagulant **NOAC NVAF** Non-valvular Atrial Fibrillation

Oral Anticoagulation OAC

 NIS Protocol
 

 BI Study Number 1160-0308
 c37044336-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

PASS Post-Authorization Safety Study

RE-LY Randomized Evaluation of Long-term Anticoagulant Therapy

ROCKET-AF The Rivaroxaban Once Daily Oral Direct Factor Xa Inhibitor Compared

with Vitamin K Antagonism for Prevention of Stroke and Embolism Trial

in Atrial Fibrillation

SAE Serious Adverse Event SD Standard Deviation

SEAP Statistical and Epidemiological Analysis Plan

SE Systemic Embolism

s-IPTW Stabilized Inverse Probability of Treatment Weighting

TIA Transient Ischemic Attack

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. RESPONSIBLE PARTIES



NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim Name of finished medicinal | | | |
| name of finished medicinal product: Pradaxa, Xarelto | | | |
| Name of active ingr<br>Dabigatran, warfar | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| Title of study: | rivaroxaban am | ong Japanese patients with no | on-valvular atrial |
| Rationale and background: | Comparative safety and effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD) Atrial fibrillation (AF) is a common cardiac arrhythmia and is associated with 15-20% of all strokes [R96-0267], [R96-0252]. Among AF patients, the prevalence of concomitant coronary artery disease (CAD) is estimated to range from 17% to 46.5% [P17-09543], which can increase the risks of major bleeding, stroke, and mortality [R21-3491]. The management of AF is complicated by the presence of concomitant CAD when co-prescription of oral anticoagulation (OAC) with antiplatelet therapy is needed. Therefore, careful considerations are necessary in choosing antithrombotic therapies to balance the bleeding risk, stroke risk, and other thrombosis risks. Non-valvular atrial fibrillation (NVAF) is a subtype of AF. The 2020 European Society of Cardiology (ESC) Guidelines recommends nonvitamin K oral anticoagulant (NOAC) treatments over warfarin for eligible oral anticoagulant-naïve NVAF patients [P21-09613]. Dabigatran and rivaroxaban are the first two NOACs approved for thromboprophylaxis of AF, which are also the two widely used NOACs in Asia. According to RE-LY and ROCKET-AF, both dabigatran and rivaroxaban have shown at least equal efficacy compared to warfarin in the prevention of stroke/systemic embolism (SE), and dabigatran 110 mg bid demonstrates superiority over warfarin in major bleeding among NVAF patients [P09-11669], [R11-4223]. Further, post hoc or subgroup analyses of the two pivotal trials indicate consistent superiority in the safety profiles of NOACs versus warfarin among NVAF patients with concomitant CAD [P12-00109]. However, the current literature lacks comparative assessment of clinical outcomes among Asian NVAF patients with CAD who are managed with warfarin, dabigatran, or rivaroxaban in routine clinical practice. Given the increased risks of major bleeding and recurrent coronary events associated with CAD | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Name of company | | | |
|---|---|---|---|
| Name of company:<br>Boehringer Ingelhein | າ | | |
| Name of finished medicinal | | | |
| product: | culcinai | | |
| Pradaxa, Xarelto | | | |
| Name of active ingr<br>Dabigatran, warfar | | | |
| | 1 | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| Research | The study aims t | o make safety and effectiven | ess comparisons between |
| question and | warfarin, dabiga | tran, and rivaroxaban in routi | ne clinical practice among |
| objectives: | Japanese NVAF | patients with concomitant C. | AD. |
| | Primary object | | |
| | _ | risk of major bleeding between | |
| | | tween rivaroxaban and warfa | rin, among Japanese |
| | NVAF patients v | with concomitant CAD. | |
| | Sagandary ahia | ativo. | |
| | Secondary objective: To compare the net clinical benefits of dabigatran vs. warfarin, and | | |
| | - | <u> </u> | |
| | concomitant CA | n vs. warfarin, among Japanese NVAF patients with nt CAD. | |
| | Concommunit CAD. | | |
| | Further objecti | ve: | |
| | | ample size can be fulfilled and | d the baseline |
| | - | re balanced between dabigatra | |
| | | stment, to compare the safety | |
| | _ | rivaroxaban among Japanese | NVAF patients with |
| | concomitant CA | D. | |
| a | | | |
| Study design: | | e a non-interventional study | |
| | _ | the in/exclusion criteria will | be selected and will be |
| | defined as 3 patie | em groups: | |
| | Group 1: new us | ers of warfarin | |
| | _ | new users of warfarin<br>new users of dabigatran | |
| | * | | |
| | Group 3. Hew us | up 3: new users of rivaroxaban | |
| | Comparative and | lyses of the study will follow | a two-step approach. In |
| | _ | primary and secondary outco | |
| | ± ' | vill be compared between Gro | - |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| N C | | | |
|---|---|---|---|
| Name of company:<br>Boehringer Ingelheir | n | | |
| Name of finished m<br>product:<br>Pradaxa, Xarelto | | | |
| Name of active ingr<br>Dabigatran, warfar | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| | respectively. Next, a sample size calculation using results from step one will be carried out to assess the of comparisons between Group 2 and Group 3. If feasible, comparisons will be made on the same outcomes as in step one. | | |
| Population: | The study period is from April 18th, 2011 to December 31 <sup>st</sup> , 2020. Patients in the Japan database during the study period will be identified based on the following in/exclusion criteria: Inclusion Criteria 1. ≥18 years of age 2. Has one year of look-back period prior to the index date (defined as the first date of prescription for dabigatran, rivaroxaban, or warfarin during the study period) 3. New users of warfarin, dabigatran, and rivaroxaban, defined as patients without historic use of any oral anticoagulants during the look-back period 4. Has at least 1 diagnosis of NVAF during the look-back period prior to or on the index date 5. Has at least 1 diagnosis of CAD during the look-back period prior to | | |
| | or experience 2. Initiate warf associated was complication 3. Underwent of thromboeml index date | | r period due to valvular AF, AF ction or mechanical r rheumatic AF or diagnosed with venous period prior to or on the |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheir | m | | |
| Name of finished m<br>product:<br>Pradaxa, Xarelto | edicinal | | |
| Name of active ingr | | | |
| Dabigatran, warfar | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| | <ul> <li>5. Prescribed with more than 2 anti-platelet drugs per prescription (triple or quadruple anti-platelet use), or prescribed with any anti-platelet injection</li> <li>6. Patients with missing or ambiguous age or sex information</li> </ul> | | |
| Variables: | Exposure: | | |
| | Initiation of dabi | abigatran, rivaroxaban, or warfarin during the study e and duration not restricted) | |
| | Primary outcom | <u>1e</u> : | |
| | <ul> <li>Fatal or non-fatal major bleeding (defined as any blood transfusion<br/>and/or any hospitalization with associated bleeding) in all three<br/>patient groups</li> </ul> | | |
| | Secondary outco | ome: | |
| | · Composite of infarction (Magastrointesting)/into (the first occ | e outcome of stroke/systemic embolism (SE)/myocardial (MI)/all-cause mortality (inpatient)/major bleeding/major | |
| | Further outcom | <u>es</u> : | |
| | · Individual co | component of the composite outcome in all three patient | |
| | | ected at baseline): | |
| | Demographic ch<br>· Age | <u>aracteristics</u> | |
| | • | er (male/female/other) | |
| | | matologic characteristics (if a | available) |
| | | OS2-VASc score | <u>,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,</u> |
| | | LED score | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished m<br>product:<br>Pradaxa, Xarelto | edicinal | | |
| Name of active ingr<br>Dabigatran, warfar | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| | Comorbidities (l | nas at least 1 diagnosis before | or on the index date |
| | during the look- | _ | |
| | · Heart fa | ilure (yes/no) | |
| | · Periphe | ral arterial disorder (yes/no) | |
| | · Hyperte | ension (yes/no) | |
| | · Diabete | s (yes/no) | |
| | · Prior str | roke/transient ischemic attack | (TIA)/SE (yes/no) |
| | · Cerebro | vascular disease (yes/no) | |
| | · Myocar | | |
| | · Acute C | Coronary Syndrome (yes/no) | |
| | · Unstabl | e angina (yes/no) | |
| | · Bleeding history (yes/no) | | |
| | · Renal dysfunction (yes/no) | | |
| | · Hepatic dysfunction (yes/no) | | |
| | · Cancers | s (yes/no) | |
| | · Peptic u | lcer disease (yes/no) | |
| | · Obesity | (yes/no) | |
| | Baseline co-med | ication (had used the drug be | fore or on the index date |
| | during the look-b | • | |
| | - | atelet drugs (include aspirin, o<br>el) (yes/no) | clopidogrel, ticagrelor, |
| | | nber of anti-platelet drugs per<br>elet, dual antiplatelet, none) | r prescription (single |
| | · Antipla | telet use duration (single antij | platelet use: 6 months to 1 |
| | | ngle antiplatelet use: 1 month | |
| | _ | iplatelet use: <1 month, dual antiplatelet use: 6 months to | |
| | _ | year, dual antiplatelet use: 1 month to 6 months, dual antiplatelet use: <1 month, none; measured from the first | |
| | antiplatelet prescription to baseline) | | |
| | _ | roidal anti-inflammatory drug | s (ves/no) |
| | | secretion inhibitors (yes/no) | , <b>,</b> |
| | | (yes/no) | |
| | | as (yes/no) | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheir | n | | |
| Name of finished m<br>product:<br>Pradaxa, Xarelto | edicinal | | |
| Name of active ingr<br>Dabigatran, warfar | | | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| | <ul> <li>Proton pump inhibitor (yes/no)</li> <li>Antihypertensive drugs (yes/no)</li> <li>Baseline medical procedures (underwent the procedure before or on the index date during the look-back period)</li> <li>Cardioversion procedures (yes/no)</li> <li>Ablation procedures (yes/no)</li> <li>Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting (yes/no)</li> </ul> | | |
| Data sources: | acute care hospi<br>Japan. The data<br>blood test result<br>data, covering n<br>years old. Each<br>(ID) to which all<br>diagnosis is cod | st databases in Japan, collectificates which account for 25% of base contains comprehensive t data, insurance claims data, more than 35 million patients, patient is assigned a specifical inpatient and outpatient datalled according to the 10th Rever f Diseases (ICD-10) codes or | of emergency hospitals in emedical record data, and pharmacy claims a 34% of whom are ≥ 65 identification number a are linked. The rision of the International |
| size: | 17000, 11000, ar CAD being respective dabigatran as the the 12-month local According to a standard deviation of the standard deviation of the standard to the | d from April 2011 to December of 4000 NVAF adult patients ectively treated with either was first OAC (defined as no his ok-back period) within the published paper based on the tion, SD) treatment duration of a ranged from 265 (263.8) to ap exposed to the treatment the same article, the major blee atient-years. In comparison, AD are more likely to fall under the HAS-BLED score, a promong AF patients, thus incressions. | with a medical history of arfarin, rivaroxaban or tory of OAC usage during database. database, the mean of different drugs among 868 (725) days, with the e longest [P20-03503]. Eding rate for AF patients AF patients with ler high or medium/high redictor of bleeding |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal | | | |
| product: | carcinai | | |
| Pradaxa, Xarelto | | | |
| Name of active ingr<br>Dabigatran, warfar | | | |
| Protocol date: | Study | Version/Revision: | Version/Revision date: |
| Frotocor date. | number: | version/Revision. | version/Revision date. |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| | the major bleed years among Ja Furthermore, produced design and the last section of the major bleeding patients should concomitant CA. For dabigatran average exposurate of 3 per 10 patients for selected and the selected and the last section of t | vs. warfarin, if the HR is assure time to be 1 year per patients with 80% power will requind 3025 patients for each armors will require a total sample or each arm. To be conservative each arm needs around the HR of rivaroxaban was time to be 1 year per patient of patient-years with 80% powers and 4845 patient of balance the baseline characters are Probability of Treatment Varefore sample loss is expected the sample loss due to IPTW inple sizes for dabigatran and an 3781 and 6056 respectively | database. databa |
| Data analysis: | Descriptive analysis will be performed for describing patient demographic and clinical characteristics. Comparative analysis for | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal | | | |
| product:<br>Pradaxa, Xarelto | | | |
| Name of active ingr | edient. | | |
| Dabigatran, warfar | | | |
| Protocol date: | Study | Version/Revision: | Version/Revision date: |
| | number: | | |
| Nov. 15th, 2021 | 1160-0308 | 1.0 | NA |
| | primary and sec groups. | condary outcomes will be con | nducted between treatment |
| | will compare t | e analysis will follow a two-s<br>the baseline characteristics | and clinical outcomes of |
| | | AC (Dabigatran, Rivaroxaban<br>ninimize potential confoun | |
| | | of the individual NOAC group using Stabilized Inverse | |
| | Weighting (s-II | PTW). Absolute standardized balance of patient characterist | l difference (ASD) will be |
| | A Cox proportional hazard regression model with the time since NOAC drug index date as the underlying timescale will be used to compute | | |
| | adjusted hazard ratios (aHRs) with 95% CIs. If substantial covariate | | |
| | imbalance between treatment group is noted, as assessed by a standardized difference >0.1, then outcome models will be further | | |
| | adjusted by cover proportional has | variates that are out of balance zards models. | e using multivariable Cox |
| | | p will determine whether the ween dabigatran and rivarox | ± |
| | - | is the required sample size | <b>O</b> 1 |
| | _ | rivaroxaban-treated groups. I<br>juirement, analysis will move | |
| | analysis betwee | n the two NOAC groups. | • |
| | For each component outcome of all 3 groups, the event-free survival will be plotted with Kaplan-Meier curves after s-IPTW adjustments. | | |
| | A sensitivity analysis will be conducted for primary and secondary outcomes by using a conventional 1:1 propensity score matching method to assess the robustness of the s-IPTW model. | | |
| Milestones: | Protocol finaliza | tion: Sep. 2021 | |
| | DMRP completi | • | |
| | Final report of st | udy results: Dec. 2021 | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|--------|------|---------------------------|---------------------|--------|
| 1 | | | | |
| 2 | | | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. MILESTONES

| Milestone | Planned Date |
|--------------------------------|--------------|
| Protocol finalization | Sep. 2021 |
| DMRP | Oct. 2021 |
| Final report of study results: | Dec. 2021 |

#### 7. RATIONALE AND BACKGROUND

Atrial fibrillation (AF) is a common cardiac arrhythmia and is associated with 15-20% of all strokes [R96-0267], [R96-0252]. Among AF patients, the prevalence of concomitant coronary artery disease (CAD) is estimated to range from 17% to 46.5% [P17-09543], which can increase the risks of major bleeding, stroke, and mortality [R21-3491]. The management of AF is complicated by the presence of concomitant CAD when co-prescription of oral anticoagulation (OAC) with antiplatelet therapy is needed. Therefore, careful considerations are necessary in choosing antithrombotic therapies to balance the bleeding risk, stroke risk, and other thrombosis risks.

Non-valvular atrial fibrillation (NVAF) is a subtype of AF. The 2020 European Society of Cardiology (ESC) Guidelines recommends non-vitamin K oral anticoagulant (NOAC) treatments over warfarin for eligible oral anticoagulant-naïve NVAF patients [P21-09613]. Dabigatran and rivaroxaban are the first two NOACs approved for thromboprophylaxis of AF, which are also the two widely used NOACs in Asia. According to RE-LY and ROCKET-AF, both dabigatran and rivaroxaban have shown at least equal efficacy compared to warfarin in the prevention of stroke/systemic embolism (SE), and dabigatran 110 mg bid demonstrates superiority over warfarin in major bleeding among NVAF patients [P09-11669], [R11-4223]. Further, post hoc or subgroup analyses of the two pivotal trials indicate consistent superiority in the safety profiles of NOACs versus warfarin among NVAF patients with concomitant CAD [P12-00109]. However, the current literature lacks comparative assessment of clinical outcomes among Asian NVAF patients with CAD who are managed with warfarin, dabigatran, or rivaroxaban in routine clinical practice. Given the increased risks of major bleeding and recurrent coronary events associated with CAD, it is necessary to evaluate the safety outcomes and net clinical benefits among Asian NVAF patients with concomitant CAD.

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. RESEARCH QUESTION AND OBJECTIVES

The study aims to make safety and effectiveness comparisons between warfarin, dabigatran, and rivaroxaban in routine clinical practice among Japanese NVAF patients with concomitant CAD.

#### **Primary objective:**

To compare the risk of major bleeding between dabigatran and warfarin, and between rivaroxaban and warfarin, among Japanese NVAF patients with concomitant CAD

#### Secondary objective:

To compare the net clinical benefits of dabigatran vs. warfarin, and rivaroxaban vs. warfarin, among Japanese NVAF patients with concomitant CAD. Specifically, the composite outcome will be used to indicate net clinical benefits.

#### **Further objective:**

If the required sample size can be fulfilled and the baseline characteristics are balanced between dabigatran and rivaroxaban groups after IPTW adjustment, to compare the safety and net clinical benefits of dabigatran vs rivaroxaban among Japanese NVAF patients with concomitant CAD.

#### 9. RESEARCH METHODS

#### 9.1 STUDY DESIGN

This study will be a non-interventional cohort study based on existing data. Patients meeting the in/exclusion criteria will be selected and will be defined as 3 patient groups:

Group 1: new users of warfarin Group 2: new users of dabigatran Group 3: new users of rivaroxaban

Comparative analyses of the study will follow a two-step approach. In the first step, the primary and secondary outcomes, as well as baseline characteristics, will be compared between Group 1&2 and Group 1&3, respectively.

The second step will utilize the estimated results from step one, which are HRs of major bleeding events between Group 1&2 and between Group 1&3 among NVAF patients with concomitant CAD, to carry out a more accurate sample size calculation to compare dabigatran versus rivaroxaban. If feasible, comparisons will be made on the same outcomes as in step one.

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2 SETTING

Study Period: the entire time period that includes the look-back period, the cohort entry date (drug index date), and follow-up period for the study population. The study period will be from April 18th, 2011 (start of data collection) to December 31st, 2020 (end of data collection).

Patient Selection Period: the time period for which patients are eligible to enter the cohort, which is from April 18th, 2012 to December 31st, 2020.

Cohort Entry Date: The drug index date, defined as the first date of prescription for dabigatran, rivaroxaban, or warfarin during the patient selection period.

Look-back Period: the 365-day period that ends 1 day prior to the cohort entry date. The earliest start date of the look-back period is April 18th, 2011.

Loss of follow-up: the last data point available in the database during the study period.

Follow-Up Period: the period starting from the cohort entry date (first prescription of the drug of interest) and ending at the earliest occurrence of the following:

- Discontinuation of the index OAC, defined as a continuous gap of 45 days or more between the expected refill date and the actual refill date (discontinuation date defined as 45 days after the expected refill date)
- Switching to another OAC, if the index OAC is discontinued and another OAC is started within 45 days of the expected refill date of the index OAC
- · Loss of follow-up
- Occurrence of outcomes of interest (for primary outcome: major bleeding; for secondary outcome: the onset of the first occurring component event; for further outcomes: the respective onset of component events)
- Death (except for analyses for the composite outcome and all-cause mortality as a component outcome)
- End of study period

The notion of enrollment is not defined in \_\_\_\_\_\_ Therefore, a proxy enrolment criterion defined as start of enrolment = date of first inpatient/outpatient encounter; end of enrolment = date of last inpatient/outpatient encounter will be used. "Enrolment" herein will refer to this proxy enrolment measure. For entry into the study population, patients will be required to have had at least 365 days of enrollment prior to the cohort entry date.

#### 9.2.1 Study Sites

The study will be based on existing data from the database, which covers all insurance types and a large population size (9.4). Thus, selection bias can be minimized.

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2.2 Study population

The target population of the study are Japanese NVAF patients with concomitant CAD, who are prescribed with dabigatran, rivaroxaban, or warfarin. The source population of the study are Japanese patients in the Japan (a) database during the study period, which is from April 18<sup>th</sup>, 2011 to December 31<sup>st</sup>, 2020. The study population will be selected based on the following in/exclusion criteria:

#### Inclusion Criteria

- 1.  $\geq$ 18 years of age
- 2. Has one year of look-back period prior to the index date (defined as the first date of prescription for dabigatran, rivaroxaban, or warfarin during the study period)
- 3. New users of warfarin, dabigatran, and rivaroxaban, defined as patients without historic use of any oral anticoagulants during the look-back period
- 4. Has at least 1 diagnosis of NVAF during the look-back period prior to or on the index date
- 5. Has at least 1 diagnosis of CAD during the look-back period prior to or on the index date

#### **Exclusion Criteria**

- 1. Diagnosed with end-stage renal disease, or undergo hemodialysis, or experience pregnancy during the study period
- 2. Initiate warfarin, dabigatran, rivaroxaban due to valvular AF, AF associated with mechanical valve malfunction or mechanical complication of heart valve prosthesis, or rheumatic AF
- 3. Underwent joint replacement procedures or diagnosed with venous thromboembolism during the look-back period prior to or on the index date
- 4. Prescribed with more than 1 OAC on the index date
- 5. Prescribed with more than 2 anti-platelet drugs per prescription (triple or quadruple antiplatelet use), or prescribed with any anti-platelet injection
- 6. Patients with missing or ambiguous age or sex information

#### 9.2.3 Study visits

This is a non-interventional study based on existing data, hence not applicable.

### 9.2.4 Study discontinuation

This is a non-interventional study based on existing data, hence not applicable.

#### 9.3 VARIABLES

#### 9.3.1 Exposures

#### Exposure:

Respectively for Group 1, 2, and 3, the initiation of warfarin, dabigatran, or rivaroxaban during the study period (dosage and duration are not restricted).

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The exposure is measured through drug prescription records, which is recorded as Receipt Code. In the database, information pertinent to exposure records include the date of dispensing, drug quantity, dose, number of days of prescription supply, and prescriber.

#### 9.3.2 Outcomes

Outcomes are recorded with the 10th Revision of the International Classification of Diseases (ICD-10) codes. In the database, information related to outcomes include the date of occurrence, the number of events, and the severity. All outcomes are incident events after the index date.

#### 9.3.2.1 Primary outcomes

#### **Primary outcome:**

• Fatal or non-fatal major bleeding (defined as any blood transfusion and/or any hospitalization with associated bleeding) in all three patient groups

#### 9.3.2.2 Secondary outcomes

#### **Secondary outcome:**

• Composite outcome of stroke/SE/MI/all-cause mortality (inpatient) /major bleeding/major GI bleeding (hospitalization due to GI bleeding)/ICH in all three patient groups (the first occurrence of any of the component events counts as an event; this outcome indicates the net clinical benefit)



#### 9.3.3 Covariates

Covariates are recorded with the 10th Revision of the International Classification of Diseases (ICD-10) codes for disease diagnosis and Receipt Code for medications.

#### **Covariates (collected at baseline):**

Demographic characteristics

- · Age
- Gender (male/female/other)

Ischemic and hematologic characteristics (if available)

- CHA2DS2-VASc score
- · HAS-BLED score

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Comorbidities (has at least 1 diagnosis before or on the index date during the look-back period)

- · Heart failure (yes/no)
- Peripheral arterial disorder (yes/no)
- Hypertension (yes/no)
- · Diabetes (yes/no)
- Prior stroke/transient ischemic attack (TIA)/SE (yes/no)
- · Cerebrovascular disease (yes/no)
- Myocardial infarction (yes/no)
- Acute Coronary Syndrome (yes/no)
- · Unstable angina (yes/no)
- Bleeding history (yes/no)
- Renal dysfunction (yes/no)
- Hepatic dysfunction (yes/no)
- · Cancers (yes/no)
- · Peptic ulcer disease (yes/no)
- · Obesity (yes/no)

# Baseline co-medication (had used the drug before or on the index date during the look-back period)

- · Anti-platelet drugs (include aspirin, clopidogrel, ticagrelor, prasugrel) (yes/no)
- The number of anti-platelet drugs per prescription (single antiplatelet, dual antiplatelet, none)
- Antiplatelet use duration (single antiplatelet use: 6 months to 1 year, single antiplatelet use: 1 month to 6 months, single antiplatelet use: <1 month, dual antiplatelet use: 6 months to 1 year, dual antiplatelet use: 1 month to 6 months, dual antiplatelet use: <1 month, none; measured from the first antiplatelet prescription to baseline)
- · Nonsteroidal anti-inflammatory drugs (yes/no)
- · Gastric secretion inhibitors (yes/no)
- · Statins (yes/no)
- · Heparins (yes/no)
- Proton pump inhibitor (yes/no)
- Antihypertensive drugs (yes/no)

# Baseline medical procedures (underwent the procedure before or on the index date during the look-back period)

- · Cardioversion procedures (yes/no)
- · Ablation procedures (yes/no)
- · Percutaneous Coronary Intervention or Coronary Artery Bypass Grafting (yes/no)

#### 9.4 DATA SOURCES

The \_\_\_\_\_\_\_) database is one of the largest databases in Japan, collecting data from over 400 acute care hospitals which account for 25% of emergency hospitals in Japan. The database contains comprehensive medical record data,

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

blood test result data, insurance claims data, and pharmacy claims data, covering more than 35 million patients, 34% of whom are  $\geq$  65 years old. Each patient is assigned a specific identification number (ID) to which all inpatient and outpatient data are linked. The diagnosis is coded according to the  $10^{th}$  Revision of the International Classification of Diseases (ICD-10) codes or local disease codes.

The distribution of demographic characteristics, including age and sex, of patients registered in the database is very similar to the distribution of these characteristics of patients visiting hospitals in Japan.

#### 9.5 STUDY SIZE

During the period from April 2011 to December 2020, there are roughly 17000, 11000, and 4000 NVAF adult patients with a medical history of CAD being respectively treated with either warfarin, rivaroxaban or dabigatran as the first OAC (defined as no history of OAC usage during the 12-month look-back period) within the database.

According to a published paper based on the database, the mean (standard deviation, SD) treatment duration of different drugs among new user groups ranged from 265 (263.8) to 868 (725) days, with the dabigatran group exposed to the treatment the longest [P20-03503]. According to the same article, the major bleeding rate for AF patients is 1.5 per 100 patient-years. In comparison, AF patients with concomitant CAD are more likely to fall under high or medium/high risk categories of the HAS-BLED score, a predictor of bleeding complications among AF patients, thus increasing the event rate for major bleeding about 2-3 times [P09-11669], [R11-4223]. Therefore, the major bleeding rate is assumed to be rather 3-4.5 per 100 patient-years among Japanese AF+CAD patients in the database. Furthermore, previous analysis concluded substantial superiority of dabigatran (HR=0.66, 95% CI 0.529-0.825) and rivaroxaban (HR=0.74, 95% CI 0.618-0.879) over warfarin in major bleeding among AF patients [P09-11669], [R11-4223]. The comparative rates of major bleeding between individual NOAC- and warfarin- treated patients should follow a similar trend among NVAF patients with concomitant CAD.

For dabigatran vs. warfarin, if the HR is assumed to be 0.66 and the average exposure time to be 1 year per patient, an event rate of 3 per 100 patient-years with 80% power will require a total sample size of 6050 patients and 3025 patients for each arm; an event rate of 4.5 per 100 patient-years will require a total sample size of 4040 patients and 2020 patients for each arm. To be conservative, the lower bound is selected and therefore each arm needs around 3025 patients.

Similarly, assuming the HR of rivaroxaban vs. warfarin is 0.74 and the average exposure time to be 1 year per patient, the lower-bound event rate of 3 per 100 patient-years with 80% power will require a total sample size of 9690 patients and 4845 patients for each arm.

Additionally, to balance the baseline characteristics between groups, truncated Inverse Probability of Treatment Weighting (IPTW) will be applied and therefore sample loss is expected. In NOAC vs. warfarin comparisons, if the sample loss due to IPTW truncation is assumed to be 20%, the sample sizes for dabigatran and rivaroxaban groups need to be greater than 3781 and 6056 respectively, which can be satisfied by the database.

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.6 DATA MANAGEMENT

The data management plan is summarized below. Full details of the data management plan are documented in a separate NIS-Data Management and Review Plan (NIS-DMRP). The data will be managed by BI. Source code of data management and data analyses will be kept for inspection at least for five years after publication of the results.

#### 9.7 DATA ANALYSIS



Descriptive analysis will be performed for describing patient demographic and clinical characteristics. For categorical variables, the frequency (n) and percentage (%) of patients under each category will be calculated. For continuous variables, the mean, median, standard deviations, interquartile range and minimum and maximum will be summarized.

In comparative analysis, the number of patients, number of events, number of person-years, incidence rate, and incidence proportion will be reported for all outcomes. Incidence rate of each outcome for each treatment group will be reported as the number of events (counts the first event per patient) divided by the total number of person-years at risk during follow-up. In addition, the incidence proportion of each outcome for each treatment group will be reported as the number of events (counts the first event per patient) divided by the total number of patients at risk.

Incidence rate of each outcome for each treatment group will be reported as the main descriptive statistics.

Table shells are attached as Annex 3.

#### 9.7.1 Main analysis

Comparative analysis for primary and secondary outcomes will be conducted between treatment groups. The comparative analysis will follow a two-step approach. The first step will compare the baseline characteristics and clinical outcomes of individual NOAC (Dabigatran, Rivaroxaban) -versus warfarin-treated groups.

During the first step of the comparative analysis, the baseline characteristics of the individual NOAC groups will be balanced with the warfarin group to account for potential confounding effects. Propensity scores will be calculated based on multinomial logistic regressions, with all covariates being incorporated. Next, an inverse probability of treatment weighting (IPTW) method will be applied using the calculated propensity score to avoid sample size inflation and to ensure appropriate estimation of variances. Yet, the IPTW estimates can be heavily influenced by large weights, thus destabilizing the results. To increase the robustness of the model, weight truncation will be applied once the distribution of propensity score is available. The distribution of propensity scores will be described, based on which the cut-off points of weight estimates will be chosen. Lastly, the calculated stabilized IPTW (s-IPTW) estimates will be applied to obtain two comparative pairs of individual NOAC vs. warfarin groups, for which the baseline demographics, risk factors, and clinical characteristics will be compared

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

using the absolute standardized difference (ASD) pre- and post- IPTW to assess the balance and model robustness. A covariate (baseline demographics, risk factors, clinical characteristics) will be considered well balanced if the ASD is below 0.1.

A Cox proportional hazard regression model with the time since NOAC drug index date as the underlying timescale will be used to compute adjusted hazard ratios (aHRs) with 95% CIs. If substantial covariate imbalance between treatment group is noted assessed by a standardized difference >0.1, then outcome models will be further adjusted by covariates that are out of balance using multivariable Cox proportional hazards models.

The second step will determine whether the patient characteristics are comparable between dabigatran and rivaroxaban treatment groups and whether there is the required sample size for comparisons between dabigatran- and rivaroxaban-treated groups. If the database can fulfil the sample size requirement, analysis will move forward for comparative analysis between the two NOAC groups.

For each component outcome of all 3 groups, the event-free survival will be plotted with Kaplan-Meier curves after s-IPTW adjustments.



#### 9.7.3 Safety Analysis

Please refer to the other analysis sections.

#### 9.8 QUALITY CONTROL

The quality control, review, and monitoring plan are summarized below. Greater details are documented in the NIS-DMRP.

The study will strictly follow BI NIS SOP, PASS SOP and any other relevant SOPs. In addition, this study will follow key elements of the Guideline for Good Pharmacoepidemiology Practices (GPP) and Good Pharmacovigilance Practice (GVP). The statistical analytic approach will be reviewed/repeated by a second analyst. The study report will be reviewed, approved and archived per BI SOP.

Whenever possible, validated algorithm will be used for variables, including exposure, outcomes, and covariates, to minimize misclassification and information bias.



## NIS Protocol BI Study Number 1160-0308

 **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Quality controls include checks for the validity and logical content of codes and checks for missing values and variables.

The Analyst from BI assigned to the study will perform a cross-review of the different tables of results.

In order to control for potential inconsistencies and errors, all variables will be tabulated. The distribution of each variable will be examined. Extreme observations with values larger than  $\pm$  3 standard deviations (SD) will be examined as potential outliers and consequently excluded from the dataset.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

This is a non-interventional study based on existing data. The data do not include vital signs or laboratory test results (e.g. blood pressure, international normalized ratio values, renal function parameters). Therefore, the study may be subject to potential residual confounding due to the absence of certain key data.

Further, the database contains around 23% of emergency care hospitals in Japan, which does not form a fully closed healthcare system and therefore could lead to information bias. Additionally, the mortality is only known for hospitalized patients during hospitalization, thus resulting in inaccurate estimates of the mortality rate.

Due to the above reasons, the study results might not be generalizable to the entire AF patient population in Japan.

#### 9.10 OTHER ASPECTS

Not Applicable.

#### 9.10.1 Data quality assurance

The quality assurance auditor will have access to the investigator's study-related files and correspondence of this study.

### 9.10.2 Study records

#### 9.10.2.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at BI.

#### 9.10.2.2 Direct access to source data and documents

All source documents must be available at all times for review by BI, IRB/IEC, auditor and inspection by health authorities.

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.10.3 Protocol deviations

The investigators or sub-investigators will not develop or implement any deviation or change to the protocol without prior review by BI.

#### 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, Guidelines for Good Pharmacoepidemiology Practice (GPP), and the relevant BI Standard Operating Procedures (SOPs).

# 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This NIS will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB)/Independent Ethics Committee (IEC) and Competent Authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

#### 10.2 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Only anonymized data will be used in the study. Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB/IEC and the regulatory authorities.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11.1 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

#### Collection of AEs

This study is a non-interventional study based on secondary data without involving review or analysis of any individual patient level data. The data is extracted and analyzed in an aggregate manner. Therefore, from safety information collecting perspective, no AE/ADR collection & reporting of individual case safety reports is required. .

#### 11.2 REPORTING TO HEALTH AUTHORITIES

Based on current guidelines from the International Society for Pharmacoepidemiology [R11-4318] and the European Medicines Agency (EMA) [R16-4913], non-interventional studies conducted using health care records do not require expedited reporting of suspected adverse events/reactions. Specifically, as stated in section VI.C.1.2.1 of GVP, Module VI – Management and Reporting of Adverse Reactions to Medicinal Products, for non-interventional study designs, which are based on use of secondary data, reporting of adverse reactions is not required.

This study is a non-interventional study based on secondary data, which will not involve individual medical record review. Therefore, no AE/ADR collection of this study will be performed and reported to Chinese regulatory authorities.

This study is classified as a PASS, and the study report will be reported to health authorities according to local regulations. The study results will also be reflected in the PSURs.

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

BI intends to use data from this study to prepare peer-reviewed publications and other scientific communications such as abstracts, posters, and podiums presentations.

The final report of the study result is planned in December 2021. Results of this PASS will be disclosed on encepp.eu and ClinicalTrials.gov.

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

[R96-0267] Wolf, P. A. (1987). Atrial fibrillation: A major contributor to stroke in the elderly. The Framingham Study. Archives of Internal Medicine, 147(9), 1561–1564. https://doi.org/10.1001/archinte.147.9.1561

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

[R96-0252] Wolf, P. A., Abbott, R. D., & Kannel, W. B. (1991). Atrial fibrillation as an independent risk factor for stroke: The Framingham Study. Stroke, 22(8), 983–988. https://doi.org/10.1161/01.str.22.8.983

[P17-09543] Michniewicz E, Mlodawska E, Lopatowska P, Tomaszuk-Kazberuk A, Malyszko J. Patients with atrial fibrillation and coronary artery disease - Double trouble. Adv Med Sci. 2018 Mar;63(1):30-35. doi: 10.1016/j.advms.2017.06.005. Epub 2017 Aug 14. PMID: 28818746.

[R21-3491] Kralev S, Schneider K, Lang S, Süselbeck T, Borggrefe M. Incidence and severity of coronary artery disease in patients with atrial fibrillation undergoing first-time coronary angiography. Plos one. 2011;6(9):e24964. DOI: 10.1371/journal.pone.0024964. PMID: 21957469; PMCID: PMC3177852.

[P21-09613] Hindricks G, Potpara T, Dagres N, Arbelo E, Bax JJ, Blomström-Lundqvist C, Boriani G, Castella M, Dan GA, Dilaveris PE, Fauchier L, Filippatos G, Kalman JM, La Meir M, Lane DA, Lebeau JP, Lettino M, Lip GYH, Pinto FJ, Thomas GN, Valgimigli M, Van Gelder IC, Van Putte BP, Watkins CL; ESC Scientific Document Group. 2020 ESC Guidelines for the diagnosis and management of atrial fibrillation developed in collaboration with the European Association for Cardio-Thoracic Surgery (EACTS): The Task Force for the diagnosis and management of atrial fibrillation of the European Society of Cardiology (ESC) Developed with the special contribution of the European Heart Rhythm Association (EHRA) of the ESC. Eur Heart J. 2021 Feb 1;42(5):373-498. doi: 10.1093/eurheartj/ehaa612. Erratum in: Eur Heart J. 2021 Feb 1;42(5):507. Erratum in: Eur Heart J. 2021 Feb 1;42(5):507. Erratum in: Eur Heart J. 2021 Sep 14;: PMID: 32860505.

[P09-11669] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. Erratum in: N Engl J Med. 2010 Nov 4;363(19):1877. PMID: 19717844.

[R11-4223] Patel MR, Mahaffey KW, Garg J, Pan G, Singer DE, Hacke W, Breithardt G, Halperin JL, Hankey GJ, Piccini JP, Becker RC, Nessel CC, Paolini JF, Berkowitz SD, Fox KA, Califf RM; ROCKET AF Investigators. Rivaroxaban versus warfarin in nonvalvular atrial fibrillation. N Engl J Med. 2011 Sep 8;365(10):883-91. doi: 10.1056/NEJMoa1009638. Epub 2011 Aug 10. PMID: 21830957.

[P12-00109] Hohnloser SH, Oldgren J, Yang S, Wallentin L, Ezekowitz M, Reilly P, Eikelboom J, Brueckmann M, Yusuf S, Connolly SJ. Myocardial ischemic events in patients with atrial fibrillation treated with dabigatran or warfarin in the RE-LY (Randomized Evaluation of Long-Term Anticoagulation Therapy) trial. Circulation. 2012 Feb 7;125(5):669-76. doi: 10.1161/CIRCULATIONAHA.111.055970. Epub 2012 Jan 3. PMID: 22215856.

[P20-03503] Kohsaka S, Katada J, Saito K, et al. Safety and effectiveness of non-vitamin K oral anticoagulants versus warfarin in real-world patients with non-valvular atrial fibrillation: a retrospective analysis of contemporary Japanese administrative claims data. Open Heart 2020;7:e001232. doi: 10.1136/openhrt-2019-001232

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

[R11-4318] ISPE. (April 2007). Guidelines for good pharmacoepidemiology practices (GPP).International Society for Pharmacoepidemiology.

http://www.pharmacoepi.org/resources/guidelines 08027.cfm (access date: 9 October 2021)

[R16-4913] European Medicines Agency (EMA). (8 September 2014). Guideline on good pharmacovigilance practices (GVP): module VI - management and reporting of adverse reactions to medicinal products (rev 1). European Medicines Agency (EMA). http://www.ema.europa.eu/docs/en\_GB/document\_library/Scientific\_guideline/2014/0 9/WC500172402.pdf (access date: 9 October 2021)

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference Number | Date | Title |
|--------|------------------------------|------|-------|
| 1 | | | |

#### ANNEX 2. ENCEPP CHECKLIST FOR STUDY PROTOCOLS

Doc.Ref. EMA/540136/2009

## **ENCePP Checklist for Study Protocols (Revision 4)**

Adopted by the ENCePP Steering Group on 15/10/2018

The European Network of Centres for Pharmacoepidemiology and Pharmacovigilance (ENCePP) welcomes innovative designs and new methods of research. This Checklist has been developed by ENCePP to stimulate consideration of important principles when designing and writing a pharmacoepidemiological or pharmacovigilance study protocol. The Checklist is intended to promote the quality of such studies, not their uniformity. The user is also referred to the ENCePP Guide on Methodological Standards in Pharmacoepidemiology, which reviews and gives direct electronic access to guidance for research in pharmacoepidemiology and pharmacovigilance.

For each question of the Checklist, the investigator should indicate whether or not it has been addressed in the study protocol. If the answer is "Yes", the section number of the protocol where this issue has been discussed should be specified. It is possible that some questions do not apply to a particular study (for example, in the case of an innovative study design). In this case, the answer 'N/A' (Not Applicable) can be checked and the "Comments" field included for each section should be used to explain why. The "Comments" field can also be used to elaborate on a "No" answer.

This Checklist should be included as an Annex by marketing authorisation holders when submitting the protocol of a non-interventional post-authorisation safety study (PASS) to a regulatory authority (see the Guidance on the format and content of the protocol of non-interventional post-authorisation safety studies). The Checklist is a supporting document and does not replace the format of the protocol for PASS presented in the Guidance and Module VIII of the Good pharmacovigilance practices (GVP).

#### Study title:

Comparative safety and effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD)

**EU PAS Register® number:** EUPAS41345

**NIS Protocol** BI Study Number 1160-0308

 c37044336-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Stud | dy reference number (if applicable): 1160-03 | 80 | | | |
|---|---|---|---|---|---|
| Sect | ion 1: Milestones | Yes | No | N/A | Section<br>Number |
| 1.1 | Does the protocol specify timelines for | | | | |
| | 1.1.1 Start of data collection <sup>1</sup> | | | | 6.0 |
| | 1.1.2 End of data collection <sup>2</sup> | | | | 6.0 |
| | 1.1.3 Progress report(s) | | | $\boxtimes$ | |
| | 1.1.4 Interim report(s) | | | | 6.0 |
| | 1.1.5 Registration in the EU PAS Register® | | | $\boxtimes$ | |
| | 1.1.6 Final report of study results. | | | | 6.0 |
| Comn | nents: | | | | |
| | | 1 | ı | | |
| Sect | tion 2: Research question | Yes | No | N/<br>A | Section<br>Number |
| 2.1 | Does the formulation of the research question and objectives clearly explain: | | | | |
| | 2.1.1 Why the study is conducted? (e.g. to address an important public health concern, a risk identified in the risk management plan, an emerging safety issue) | | | | 7.0 |
| | 2.1.2 The objective(s) of the study? | | | | 8.0 |
| | 2.1.3 The target population? (i.e. population or subgroup to whom the study results are intended to be generalised) | | | | 9.2.2 |
| | 2.1.4 Which hypothesis(-es) is (are) to be tested? | | | $\boxtimes$ | 8.0 |
| | 2.1.5 If applicable, that there is no <i>a priori</i> hypothesis? | | $\boxtimes$ | | 8.0 |
| Comn | nents: | | | | |
| Sect | tion 3: Study design | Yes | No | N/<br>A | Section<br>Number |
| 3.1 | Is the study design described? (e.g. cohort, case-control, cross-sectional, other design) | | | | 9.1 |
| 3.2 | Does the protocol specify whether the study is based on primary, secondary or combined data collection? | | | | 9.1 |
| 3.3 | Does the protocol specify measures of | | | | 9.3.2 |

occurrence? (e.g., rate, risk, prevalence)

<sup>&</sup>lt;sup>1</sup> Date from which information on the first study is first recorded in the study dataset or, in the case of secondary use of data, the date from which data extraction starts.

Date from which the analytical dataset is completely available.

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| Sect | ion 3: Study design | Yes | No | N/<br>A | Section<br>Number |
|---|---|---|---|---|---|
| 3.4 | Does the protocol specify measure(s) of association? (e.g. risk, odds ratio, excess risk, rate ratio, hazard ratio, risk/rate difference, number needed to harm (NNH)) | $\boxtimes$ | | | 9.7 |
| 3.5 | Does the protocol describe the approach for the collection and reporting of adverse events/adverse reactions? (e.g. adverse events that will not be collected in case of primary data collection) | | | | 11.0 |
| Comm | nents: | | | | |
| Sect | ion 4: Source and study populations | Yes | No | N/<br>A | Section<br>Number |
| 4.1 | Is the source population described? | | | | 9.4 |
| 4.2 | Is the planned study population defined in terms of: | | | | |
| | 4.2.1 Study time period | $\boxtimes$ | | | 9.2.2 |
| | 4.2.2 Age and sex | $\boxtimes$ | | | 9.2.2 |
| | 4.2.3 Country of origin | $\boxtimes$ | | | 9.2.2 |
| | 4.2.4 Disease/indication | $\boxtimes$ | | | 9.2.2 |
| | 4.2.5 Duration of follow-up | | | | 9.2.2 |
| 4.3 | Does the protocol define how the study population will be sampled from the source population? (e.g. event or inclusion/exclusion criteria) | | | | 9.2.2 |
| Comm | nents: | | | | |
| | ion 5: Exposure definition and surement | Yes | No | N/<br>A | Section<br>Number |
| 5.1 | Does the protocol describe how the study exposure is defined and measured? (e.g. operational details for defining and categorising exposure, measurement of dose and duration of drug exposure) | | | | 9.3.1 |
| 5.2 | Does the protocol address the validity of the exposure measurement? (e.g. precision, accuracy, use of validation sub-study) | | | | |
| 5.3 | Is exposure categorised according to time windows? | | | | |
| 5.4 | Is intensity of exposure addressed? (e.g. dose, duration) | $\boxtimes$ | | | 9.3.1 |
| 5.5 | Is exposure categorised based on biological mechanism of action and taking into account the pharmacokinetics and pharmacodynamics of the drug? | | | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| | ion 5: Exposure definition and surement | Yes | No | N/<br>A | Section<br>Number |
|---|---|---|---|---|---|
| 5.6 | Is (are) (an) appropriate comparator(s) identified? | | | | 9.1 |
| Comm | nents: | | | | |
| | ion 6: Outcome definition and surement | Yes | No | N/<br>A | Section<br>Number |
| 6.1 | Does the protocol specify the primary and secondary (if applicable) outcome(s) to be investigated? | | | | 9.3.2 |
| 6.2 | Does the protocol describe how the outcomes are defined and measured? | | | | 9.3.2 |
| 6.3 | Does the protocol address the validity of outcome measurement? (e.g. precision, accuracy, sensitivity, specificity, positive predictive value, use of validation sub-study) | | $\boxtimes$ | | |
| 6.4 | Does the protocol describe specific outcomes relevant for Health Technology Assessment? (e.g. HRQoL, QALYS, DALYS, health care services utilisation, burden of disease or treatment, compliance, disease management) | | | | |
| Comn | nents: | | | | |
| Sect | ion 7: Bias | Yes | No | N/<br>A | Section<br>Number |
| 7.1 | Does the protocol address ways to measure | | | | Number |
| | confounding? (e.g. confounding by indication) | $\boxtimes$ | | | 9.7.1 |
| 7.2 | | | | | |
| 7.2 | confounding? (e.g. confounding by indication) Does the protocol address selection bias? (e.g. | | | | |
| 7.3 | confounding? (e.g. confounding by indication) Does the protocol address selection bias? (e.g. healthy user/adherer bias) Does the protocol address information bias? (e.g. misclassification of exposure and outcomes, time- | | | | 9.7.1 |
| 7.3 | confounding? (e.g. confounding by indication) Does the protocol address selection bias? (e.g. healthy user/adherer bias) Does the protocol address information bias? (e.g. misclassification of exposure and outcomes, time-related bias) | | | | 9.7.1 |
| 7.3<br>Comm | confounding? (e.g. confounding by indication) Does the protocol address selection bias? (e.g. healthy user/adherer bias) Does the protocol address information bias? (e.g. misclassification of exposure and outcomes, time-related bias) | | □ | N/A | 9.7.1 |
| 7.3<br>Comm | confounding? (e.g. confounding by indication) Does the protocol address selection bias? (e.g. healthy user/adherer bias) Does the protocol address information bias? (e.g. misclassification of exposure and outcomes, timerelated bias) ments: | | | N/A | 9.7.1<br>9.8<br>Section |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| <u>Sect</u> | ion 9: Data sources | Yes | No | N/<br>A | Section<br>Number |
|---|---|---|---|---|---|
| 9.1 | Does the protocol describe the data source(s) used in the study for the ascertainment of: | | | | |
| | 9.1.1 Exposure? (e.g. pharmacy dispensing, general practice prescribing, claims data, self-report, face-to-face interview) | $\boxtimes$ | | | 9.4 |
| | 9.1.2 Outcomes? (e.g. clinical records, laboratory<br>markers or values, claims data, self-report, patient<br>interview including scales and questionnaires, vital<br>statistics) | | | | 9.4 |
| | 9.1.3 Covariates and other characteristics? | | | | 9.4 |
| 9.2 | Does the protocol describe the information available from the data source(s) on: | | | | |
| | 9.2.1 Exposure? (e.g. date of dispensing, drug<br>quantity, dose, number of days of supply prescription,<br>daily dosage, prescriber) | | | | 9.3.1 |
| | 9.2.2 Outcomes? (e.g. date of occurrence, multiple event, severity measures related to event) | | | | 9.3.2 |
| | 9.2.3 Covariates and other characteristics? (e.g. age, sex, clinical and drug use history, comorbidity, co-medications, lifestyle) | | | | 9.3.3 |
| 9.3 | Is a coding system described for: | | | | |
| | 9.3.1 Exposure? (e.g. WHO Drug Dictionary, Anatomical Therapeutic Chemical (ATC) Classification System) | $\boxtimes$ | | | 9.3.1 |
| | 9.3.2 Outcomes? (e.g. International Classification of Diseases (ICD), Medical Dictionary for Regulatory Activities (MedDRA)) | | | | 9.3.2 |
| | 9.3.3 Covariates and other characteristics? | | | | 9.3.3 |
| 9.4 | Is a linkage method between data sources described? (e.g. based on a unique identifier or other) | | | | 9.4 |
| Comm | ients: | | | | |
| Sect | ion 10: Analysis plan | Yes | No | N/<br>A | Section<br>Number |
| 10.1 | Are the statistical methods and the reason for their choice described? | | | | 9.7 |
| 10.2 | Is study size and/or statistical precision estimated? | $\boxtimes$ | | | 9.5 |
| 10.3 | Are descriptive analyses included? | | | | 9.7 |
| 10.4 | Are stratified analyses included? | | $\boxtimes$ | | |
| 10.5 | Does the plan describe methods for analytic control of confounding? | | | | 9.7 |
| 10.6 | Does the plan describe methods for analytic control of outcome misclassification? | | $\boxtimes$ | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| T | | | I | |
|---|---|---|---|---|
| Section 10: Analysis plan | Yes | No | N/<br>A | Section<br>Number |
| 10.7 Does the plan describe methods for handling missing data? | | $\boxtimes$ | | |
| 10.8 Are relevant sensitivity analyses described? | $\boxtimes$ | | | 9.7.2 |
| Comments: | | | | |
| Section 11: Data management and quality control | Yes | No | N/<br>A | Section<br>Number |
| 11.1 Does the protocol provide information on data storage? (e.g. software and IT environment, database maintenance and anti-fraud protection, archiving) | | | | 9.6 |
| 11.2 Are methods of quality assurance described? | $\boxtimes$ | | | 9.10.1 |
| 11.3 Is there a system in place for independent review of study results? | | | | |
| Comments: | | | | |
| [ | | | | |
| Section 12: Limitations | Yes | No | N/<br>A | Section<br>Number |
| 12.1 Does the protocol discuss the impact on the study results of: | | | | |
| 12.1.1 Selection bias? | $\boxtimes$ | | | 9.9 |
| 12.1.2 Information bias? | $\boxtimes$ | | | 9.9 |
| 12.1.3 Residual/unmeasured confounding? (e.g. anticipated direction and magnitude of such biases, validation sub-study, use of validation and external data, analytical methods). | | | | 9.9 |
| 12.2 Does the protocol discuss study feasibility? (e.g. study size, anticipated exposure uptake, duration of follow-up in a cohort study, patient recruitment, precision of the estimates) | | | | 9.5 |
| Comments: | | | | |
| Section 13: Ethical/data protection issues | Yes | No | N/<br>A | Section<br>Number |
| 13.1 Have requirements of Ethics Committee/<br>Institutional Review Board been described? | $\boxtimes$ | | | 10.1 |
| 13.2 Has any outcome of an ethical review procedure been addressed? | | | | |
| 13.3 Have data protection requirements been described? | $\boxtimes$ | | | 10.2 |

**NIS Protocol** 

BI Study Number 1160-0308

 c37044336-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Section 14: Amendments and deviations | Yes | No | N/<br>A | Section<br>Number |
|---|---|---|---|---|
| 14.1 Does the protocol include a section to document amendments and deviations? | $\boxtimes$ | | | 5.0 |
| Comments: | 11 | | | |
| Section 15: Plans for communication of study | Yes | No | N/ | Section |
| results | 165 | 140 | A | Number |
| 15.1 Are plans described for communicating study results (e.g. to regulatory authorities)? | | | | 12.0 |
| 15.2 Are plans described for disseminating study results externally, including publication? | $\boxtimes$ | | | 12.0 |
| Comments: | | | hi ch | |
| 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | | |
| Name of the main author of the protocol: Date: 2021/11/15 | | | | |

#### ANNEX 3. TABLE SHELLS

Note: Table 1, Table 2a, and Table 3 are shown here to exemplify; please find the complete table shells in the attached excel file below:



Safety comparisons betv

Table 1. Patient Flow Diagram

| | Exclude<br>d | Total |
|---|---|---|
| Total number of patients MDV database 2008-04-01 - 2020-12-31 | | |
| Total number of patients MDV database in study period 2011-04-01 - 2020-12-31 | | |
| Patients prescribed with Dabigatran, or Rivaroxaban or Warfarin | | |

## NIS Protocol BI Study Number 1160-0308

 **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Patients older than 18 year old at drug index date | |
|---|---|
| Have 1y look-back prior drug index date | |
| New user of Dabigatran or Rivaroxaban or Warfarin | |
| Have at least 1 diagnosis of NVAF during the look-back period prior to or on the index date | |
| Have at least 1 diagnosis of CAD during the look-back period prior to or on the index date | |
| Excluded because of Diagnosis of end-stage renal disease, or undergo hemodialysis, or experience pregnancy during the study period | |
| Excluded because of Initiation of warfarin, dabigatran, rivaroxaban due to valvular AF, AF associated with mechanical valve malfunction or mechanical complication of heart valve prosthesis, or rheumatic AF | |
| Excluded because of Prescription with more than 1 OAC on the index date | |
| Final cohort | - |
| Warfarin | - |
| Dabigatran | - |
| Rivaroxaban | - |

Table 2a. Baseline Characteristics Comparisons – Dabigatran vs. Warfarin

| | | Overall | | s-IPTW | 'Adjust | ted | PS | PS-matched | |
|---|---|---|---|---|---|---|---|---|---|
| Variable | Da<br>big<br>atr<br>an | Warfari<br>n | Abs.<br>Std.<br>Dif | Dabigatra<br>n | Wa<br>rfar<br>in | Abs.St<br>d.Dif | Dabig<br>atran | Warf<br>arin | Abs.St<br>d.Dif |
| Age | | | | | | | | | |
| mean (sd) | | | | | | | | | |
| median [IQR] | | | | | | | | | |
| ···Min-Max | | | | | | | | | |
| Gender | | | | | | | | | |
| 1 - Male; n<br>(%) | | | | | | | | | |
| 2 - Female;<br>n (%) | | | | | | | | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| CHA2DS2-<br>VASc score |
|---|
| mean (sd) |
| median<br>[IQR] |
| ···Min-Max |
| HAS-BLED score |
| ···mean(sd) |
| ···median[IQR<br>] |
| ···Min-Max |
| Heart failure;<br>n (%) |
| Peripheral<br>arterial<br>disorder; n<br>(%) |
| Hypertension;<br>n (%) |
| Diabetes; n<br>(%) |
| Prior<br>stroke/transie<br>nt ischemic<br>attack<br>(TIA)/SE; n<br>(%) |
| Myocardial infarction; n (%) |
| Acute<br>Coronary<br>Syndrome; n<br>(%) |
| Unstable angina; n (%) |
| Bleeding<br>history; n (%) |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| • | | • | |
|---|---|---|---|
| Renal<br>dysfunction; n<br>(%) | | | |
| Hepatic<br>dysfunction; n<br>(%) | | | |
| Cancers; n (%) | <br> | | <br> |
| Peptic ulcer<br>disease; n (%) | | | |
| Cerebrovascul<br>ar disease; n<br>(%) | | | |
| Obesity; n (%) | | | |
| Anti-platelet drugs (include aspirin, clopidogrel, ticagrelor, prasugrel); n (%) | | | |
| The number of anti-platelet drugs per prescription (single antiplatelet, dual antiplatelet, none) | | | |
| single<br>antiplatelet;<br>n (%) | | | |
| dual<br>antiplatelet;<br>n (%) | | | |
| none; n (%) | | | |
| Antiplatelet use duration | | | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

| | 1 |
|---|---|
| Single<br>antiplatelet<br>use: 6<br>months to 1<br>year; n (%) | |
| Single<br>antiplatelet<br>use: 1 month<br>to 6 months;<br>n (%) | |
| Single<br>antiplatelet<br>use: <1<br>month; n (%) | |
| Dual<br>antiplatelet<br>use: 6<br>months to 1<br>year; n (%) | |
| Dual<br>antiplatelet<br>use: 1 month<br>to 6 months;<br>n (%) | |
| Dual<br>antiplatelet<br>use: <1<br>month; n (%) | |
| None; n<br>(%) | |
| Nonsteroidal<br>anti-<br>inflammator<br>y drugs; n (%) | |
| Gastric<br>secretion<br>inhibitors; n<br>(%) | |
| Statins; n (%) | |

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Heparins; n (%) |
|---|
| Proton<br>pump<br>inhibitor; n<br>(%) |
| Antihyperten<br>sive drugs; n<br>(%) |
| Cardioversio<br>n<br>procedures;<br>n (%) |
| Ablation procedures; n (%) |
| Percutaneou<br>s Coronary<br>Intervention<br>or Coronary<br>Artery<br>Bypass<br>Grafting; n<br>(%) |

Table 3. Rates and Risks of Fatal/Non-fatal Major Bleeding

| | Comparison 1 | | Comparison 2 | | Comp | arison 3* |
|---|---|---|---|---|---|---|
| | Dabig<br>atran | Warfa<br>rin | Rivaro<br>xaban | Warfa<br>rin | Dabig<br>atran | Rivaroxab<br>an |
| Rate | | | | | | |
| Overall | | | | | | |
| Number of patients | | | | | | |
| Number of events | | | | | | |
| Number of person-years | | | | | | |
| Incidence Rate per 1,000 person-<br>years (95% CI) | | | | | | |
| Incidence Proportion (n (%)) | | | | | | |
| s-IPTW adjusted | | | | | | |

NIS Protocol BI Study Number 1160-0308  c37044336-01

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Number of patients |
|----------------------------------------------------|
| Number of events |
| Number of person-years |
| Incidence Rate per 1,000 person-<br>years (95% CI) |
| Incidence Proportion (n (%)) |
| PS-matched |
| Number of patients |
| Number of events |
| Number of person-years |
| Incidence Rate per 1,000 person-<br>years (95% CI) |
| Incidence Proportion (n (%)) |
| Hazard ratios |
| s-IPTWAdjusted Hazard Ratio (95% CI) |
| PS Matched Hazard Ratio (95% CI) |

\*Note: comparison 3 will be conducted if sample size is sufficient (see section 9.5 of protocol) Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS Protocol must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI<br>product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi | X | X | X |
| Global TMM / TMMA / TM Market<br>Access | X | X | |
| Global Project Statistician | X | X | |
| Global TM RA | X | | |
| Global PVWG Chair | X | | |
| GPV SC | X | X | X |
| Global CTIS representative | X | | |
| Local Medical Director | X (if local study) | | X |
| Local Head MAcc / HEOR Director | X (if local study) | | X |
| Global TA Head Epi* | X | X | |
| Global TA Head Clinical<br>Development / Medical Affairs /<br>Market Access* | X | X | |
| Global TA Head PV RM* | X | | |
| RWE CoE | X | X | |
| PSTAT / PSTAT-MA<br>(for NISnd only) | X | X | X |
| NIS DM | X | X | X |
| Local Head MA/Clinical<br>Development | | | X (does not apply to<br>NISed without chart<br>abstraction) |

<sup>\*</sup> After review by Global TM for function

**Study Title:** Comparative safety and effectiveness of warfarin, dabigatran, and rivaroxaban among Japanese patients with non-valvular atrial fibrillation (NVAF) and concomitant coronary artery disease (CAD)

**Study Number: 1199.0308** 

Protocol Version: V1.0

NIS Protocol BI Study Number 1160-0308  **c37044336-01** 

Proprietary confidential information © 2021 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# I herewith certify that I agree to the content of the study protocol and to all documents referenced in the study protocol.

| Position: | Name/Date: | Signature: |
|-----------|------------|------------|
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |
| Position: | Name/Date: | Signature: |